CLINICAL TRIAL: NCT06309238
Title: Intensive Weight Loss Intervention Versus Bariatric Surgery for Adults With Severe and Complex Obesity: the LightBAR Randomised Trial. Lighthouse Consortium on Obesity Management (LightCOM) Trial no 4
Brief Title: Intensive Weight Loss Intervention Versus Bariatric Surgery for Adults With Severe and Complex Obesity: the LightBAR Randomised Trial
Acronym: LightBAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carsten Dirksen (Other)
Collaborators: University of Copenhagen (Other); University of Southern Denmark (Other); University of Oxford (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Responsible Party: Sponsor-Investigator, Carsten Dirksen, Associate Professor, Copenhagen University Hospital, Hvidovre
Organization: Copenhagen University Hospital, Hvidovre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LightBAR
Record Dates: First submitted 2024-02-05; First posted 2024-03-13 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the interventions, it will not be possible to blind the participants or the healthcare providers administering the interventions.
  Blinded outcome assessment will be employed for the primary outcome and anywhere else possible. When assessing clinical outcomes, the participants will be asked not to disclose their assigned intervention group to the outcome assessor. Further, they will be provided with a plain white t-shirt, or similar, to wear during clinical assessments to cover the presence of surgical scars.
  Statisticians and investigators drawing conclusions will be fully blinded. We will conduct the statistical analyses with the intervention groups coded as e.g., 'A' and 'B'. We will write two abstracts while the blinding is intact; one assuming the experimental intervention group is 'A' and the control intervention group is 'B', and one assuming the opposite. After these two abstracts have both obtained consensus, the code will be broken by the data manager.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive weight loss intervention (Experimental): The intensive weight loss intervention (IWL) includes total dietary replacements, behavioural support, and weight loss medication. The intervention consists of three phases: induction, weight loss continuation, maintenance, and it will lasts two years in total.
  Interventions: Behavioral: Intensive weight loss intervention
- Bariatric surgery (Active Comparator): Bariatric surgery: Roux-en-Y Gastric Bypass (RYGB) or Sleeve Gastrectomy (SG)
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Behavioral: Intensive weight loss intervention — Intensive weight loss intervention, incl. total meal replacements, behavioural support, and weight loss medication
  Arms: Intensive weight loss intervention
Procedure: Bariatric surgery — Roux-en-Y Gastric Bypass (RYGB) or Sleeve Gastrectomy (SG)
  Arms: Bariatric surgery

SUMMARY:
With this trial, the aim is to assess the benefits and harms of a non-surgical intensive weight loss intervention that includes total dietary replacements, behavioural support and weight-loss medication compared with bariatric surgery for people with severe and complex obesity. The interpretation of the results will help inform future care pathways for people with obesity in whom bariatric surgery is currently the only available effective treatment option.

DETAILED DESCRIPTION:
In the LightBAR trial, an intensive weight loss (IWL) intervention will be compared with bariatric surgery. The IWL consists of three phases:

'Induction' phase (week 0-12 after randomisation): total dietary replacement (TDR) programme and behavioural support with weight loss medication (WLM) if rate of weight loss is insufficient.

'Weight loss continuation' phase (week 13-32 after randomisation): progression of dietary programme including reduction in use of TDR products, reintroduction of healthy foods, with behavioural support, introduction of physical activity, WLM (as required).

'Maintenance' phase (week 33-104 after randomisation): Continued healthy diet and physical activity with WLM (if required), with return to induction phase if weight regain occurs induction, weight loss continuation, maintenance. The IWL lasts two years, and includes total dietary replacements, behavioural support, and weight loss medication. Bariatric surgery will be standard Roux-en-Y gastric bypass or sleeve gastrectomy.

ELIGIBILITY:
Please note that participants need to be invited in order to take part in the trial.

Inclusion Criteria:

* Aged 18 to 60 years (inclusive) at time of screening.
* Eligible for and willing to undergo bariatric surgery, i.e., fulfilment of criteria for bariatric surgery from the respective national health authorities:

  * DK: BMI ≥ 35 kg/m2 with one or more of the following: T2D, severe hypertension, sleep apnoea requiring treatment, symptomatic arthrosis in lower extremities, female infertility related to overweight, or BMI>40 kg/m2 with other strong medical reasons for weight loss (28). Prior to surgery, an 8% weight loss is required as well as smoking cessation.
  * UK: BMI of 35 kg/m2 to 40 kg/m2 and other significant disease (e.g., type 2 diabetes or high blood pressure), or BMI ≥40 kg/m2. Has been or is willing to receive intensive management in a specialist tier 3 obesity service (29).
* Fit for anaesthesia and surgery.
* Informed consent.

Exclusion Criteria:

* Prior bariatric or hiatal surgery, not including intragastric balloons or duodenal-jejunal bypass sleeve (Endobarrier™ or similar) if the device has been removed >1 year before screening.
* Use of any WLM (including liraglutide and semaglutide for diabetes) within last 3 months.
* Conditions that contraindicate or complicate total diet replacement (including type 1 diabetes or other diabetes requiring basal bolus insulin therapy or insulin pump therapy (for Denmark) and any diabetes requiring insulin therapy (for UK), phenylketonuria, or other conditions requiring strict adherence to special diets).
* Conditions that contraindicate or complicate treatment with GLP-1 receptor analogues (including history of pancreatitis or known allergies).
* Conditions that contraindicate or complicate bariatric surgery (GI motility disorders, large abdominal wall hernia, large hiatus hernia (>5cm), Crohn's disease, liver cirrhosis, or other conditions preventing laparoscopic bariatric surgery e.g. multiple previous abdominal surgery).
* Conditions that contraindicate or complicate study adherence and bariatric surgery (mental disorder, unstable psychiatric disease, recent history of alcohol/medication abuse, cancer treatment within 5 years).
* Pregnant or planning pregnancy in the next two years or currently breast feeding.
* Not achieving a 5% weight loss within 12 weeks prior to randomisation.
* People taking part in other research involving multidisciplinary obesity treatment that would compromise their participation in this trial.
* Another member of the household enrolled in the trial.
* Diagnosis of or treatment for severe eating disorder within the last 6 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2048-12 (Estimated)

PRIMARY OUTCOMES:
MetS-Z | 104 weeks after randomisation
  Metabolic syndrome severity Z-score

SECONDARY OUTCOMES:
Weight | 104 weeks after randomisation
  Weight (kg)
Gait speed | 104 weeks after randomisation
  4-metre gait speed (m/s)
Short-Form-36, mental component score | 104 weeks after randomisation
  Quality of life, SF36-mental component score (scale from 0-100, higher scores indicate better mental health)

OTHER OUTCOMES:
SAE | 104 weeks after randomisation
  Proportion of participants with at least one serious adverse event (according to ICH-GCP guidelines)
Proportion of participants with at least one adverse events (AE) of special interest. Each of the AE will also be assessed individually exploratorily. | 104 weeks after randomisation
  1. Anaemia (haemoglobin <6.8 mmol/L (<110 g/L))
  2. Severe and persistent/recurrent gastrointestinal symptoms (i.e.: reflux, nausea/vomiting, constipation, diarrhoea, abdominal pain - defined according to a modification of Rome IV criteria).
  3. Symptomatic hypotension (episode with loss of consciousness, seizures, or other severe mental impairments due to suspected orthostatic hypotension).
  4. Hypoglycaemia (episode with loss of consciousness, seizures or other severe mental impairments requiring third party assistance (level 3) or documented glucose concentration <3.0 mmol/l (level 2) or initiation of medication related to documented reactive hypoglycaemia).
  5. Incident alcohol abuse, other addictive disorder, self-inflicted harm, or eating disorders (Initiation of treatment (behavioural or pharmacological) for addictive disorders or documented self-inflicted harm not requiring hospitalisation (outpatient visits to emergency rooms, GP etc).
Cardiometabolic health - metabolic syndrome | 104 weeks after randomisation
  Proportion of participants with metabolic syndrome
Cardiometabolic health - blood pressure | 104 weeks after randomisation
  Systolic and diastolic blood pressure (mmHg)
Cardiometabolic health - pulse | 104 weeks after randomisation
  Pulse rate (beats per minute)
Cardiometabolic health - glucose | 104 weeks after randomisation
  Fasting glucose concentration (mmol/l)
Cardiometabolic health - Hb1Ac | 104 weeks after randomisation
  Haemoglobin A1c (mmol/mol)
Cardiometabolic health - insulin | 104 weeks after randomisation
  Fasting insulin concentration (pmol/L)
Cardiometabolic health - HOMA2-IR | 104 weeks after randomisation
  HOMA2-IR (calculated from glucose and C-peptide concentration) (ratio)
Cardiometabolic health - lipids | 104 weeks after randomisation
  Fasting lipid profile (HDL, LDL and triglycerides) (mmol/L)
Cardiometabolic health - eGFR | 104 weeks after randomisation
  Estimated Glomerular Filtration Rate (eGFR), creatinine (µmol/L), calculated from creatinine, sex and years
Cardiometabolic health - hsCRP | 104 weeks after randomisation
  High-sensitivity C-reactive protein (hsCRP), mg/L
Cardiometabolic health - Fib-4 | 104 weeks after randomisation
  Fib-4 (ALT/AST/platelets) (ratio)
Cardiometabolic health - proteinuria | 104 weeks after randomisation
  Proteinuria, measured as urine albumin/creatinine (ratio)
Cardiometabolic health - TSH | 104 weeks after randomisation
  Thyroid-stimulating hormone (IU/L)
Weight and body composition - weight loss | 104 weeks after randomisation
  Proportion of participants with body weight loss of ≥20% and ≥15%
Weight and body composition - waist circumference | 104 weeks after randomisation
  Waist circumference (cm)
Weight and body composition - body fat and lean body mass | 104 weeks after randomisation
  Body fat (%) and lean body mass (%) assessed by DXA
Physical functioning - sedentary and active | 104 weeks after randomisation
  Time spent sedentary and active (moderate to vigorous physical activity) estimated by SENS activity tracker (minutes/day)
Physical functioning - sit to stand test | 104 weeks after randomisation
  Number of sit to stands completed 30 Second Sit to Stand test
Medication use | 104 weeks after randomisation
  1. Glucose-lowering medications (number, type)
  2. Lipid-lowering medications (number, type)
  3. Blood pressure-lowering medications (number, type)
  4. Medication for pain relief (number, type)
  5. Weight loss medication (number, type)
  6. Medication used for psychiatric disorders (antidepressants, anxiolytics, antipsychotics) (number, type)
Micronutrient status, assessed as proportion of participants with deficiency | During follow-up until 104 weeks after randomisation
  1. Iron
  2. B12
  3. Folate
  4. Vitamin D
  5. Hyperparathyroidism
Bone mineral density (BMD) assessed by DXA | 104 weeks after randomisation
  1. BMD of weight bearing regions: hip (total hip and femoral neck) and lumbar region
  2. BMD of non-weight bearing region: forearm of non-dominant hand (ultradistal and 1/3 distal radius)
Sleep - ESS | 104 weeks after randomisation
  Epworth Sleepiness Scale Questionnaire Score (scale from 0-24, higher scores indicate more sleepiness)
Sleep - sleep and wake time | 104 weeks after randomisation
  Estimated sleep and wake time (minutes/day)
Sleep - sleep movement | 104 weeks after randomisation
  Movement during sleep estimated by SENS.
Health-related quality of life and mental health - EQ-5D-5L, index score | 104 weeks after randomisation
  EQ-5D-5L, index score (score between -1 and 1, higher scores indicate better health)
Health-related quality of life and mental health - EQ-5D-5L, VAS | 104 weeks after randomisation
  EQ-5D-5L, VAS score (scale from 0-100, higher scores indicate better health)
Health-related quality of life and mental health - SF-36 | 104 weeks after randomisation
  Short-Form-36, physical component score (scale from 0-100, higher scores indicate better physical health)
Health-related quality of life and mental health - EDE-Q | 104 weeks after randomisation
  Eating Disorder Examination Questionnaire (EDE-Q) score (scale from 0 to 6, higher scores indicate higher degree of eating disorder)
Health-related quality of life and mental health - WBIS-M | 104 weeks after randomisation
  Weight Bias Internalization Scale (WBIS-M) score (scale from 1-7, higher scores indicate higher degree of internalised weight bias)
Health-related quality of life and mental health - MDI | 104 weeks after randomisation
  Major Depression Inventory (MDI) (scale from 0-50, higher scores indicate more symptoms of depression)
Labour market attachment - WPAI | 104 weeks after randomisation
  Work productivity and impairment (WPAI) score points (scale from 0-100, higher scores indicate more limitations in ability to work and lower productivity)
Labour market attachment - days of sick leave | 104 weeks after randomisation
  Self-reported number of days sick leave during follow-up
Continuous glucose monitoring - hypoglycaemic range | 104 weeks after randomisation:
  Time spent in level 1 hypoglycaemic range (interstitial fluid glucose (IFG) <3.9 mmol/L)
Continuous glucose monitoring - hypoglycaemic events | 104 weeks after randomisation:
  Number of hypoglycaemic events (15 minutes of IFG<3 mmol/L)
Continuous glucose monitoring - glucose variability | 104 weeks after randomisation:
  Glucose variability (CV)
Continuous glucose monitoring - hypoglycaemic symptoms | 104 weeks after randomisation:
  Self-reported hypoglycaemic symptoms as recorded in hypoglycaemic symptom diary (reported descriptively)
Pending additional funding: Genetic profiles' (using comprehensive genetic mapping) association with the metabolic and/or weight loss response to IWL vs bariatric surgery | 104 weeks after randomisation
  1. Common gene variants with low to moderate effect on the phenotype for the construction of aggregate genetic risk scores
  2. Rare variants with potential functional effects in genes known to harbour high-impact obesity variants e.g. MC4R, LEP, LEPR, POMC, PCSK1, SIM1, NTRK2, MC3R, MRAP2, BDNF, SH2B1, KSR2
Health economy: Within-trial cost-effectiveness analysis - quality of life | 104 weeks after randomisation
  Quality of life (measured using EQ-5D-5L)
Health economy: Within-trial cost-effectiveness analysis - costs | 104 weeks after randomisation
  24-month costs, DKK
Health economy: Within-trial cost-effectiveness analysis - QALY | 104 weeks after randomisation
  Incremental cost per quality-adjusted-life-year (QALY) gained, DKK
Health economy: Model-based cost-effectiveness analysis - QALY | 104 weeks after randomisation
  Predicted lifetime QALYs gained
Health economy: Model-based cost-effectiveness analysis - healthcare costs | 104 weeks after randomisation
  Predicted lifetime healthcare costs, DKK
Health economy: Model-based cost-effectiveness analysis - cost effectiveness ratios | 104 weeks after randomisation
  Long-term incremental cost effectiveness ratios
Long-term effects - mortality and major cardiovascular disease (CVD) | 5, 10 and 20 years after randomisation
  1. Proportion of participants who die from any cause
  2. Proportion of participants with a major CVD outcome consisting of any of the following (each of the components will be assessed exploratively): myocardial infarction, stroke, hospitalisation for angina, coronary-artery bypass grafting, percutaneous coronary intervention, hospitalisation for heart failure, peripheral vascular disease
Long-term effects - prescription patterns | 5, 10 and 20 years after randomisation
  1. Proportion of participants on glucose-lowering medications
  2. Proportion of participants on lipid-lowering medications
  3. Proportion of participants on blood pressure-lowering medications
  4. Proportion of participants on medication for pain relief
  5. Proportion of participants on weight loss medication
  6. Proportion of participants on medication used for psychiatric disorders (antidepressants, anxiolytics, antipsychotics)
Long-term effect - incident cancer | 5, 10 and 20 years after randomisation
  1. Proportion of participants with any diagnosis of cancer
  2. Proportion of participants with cancers known to be associated with obesity: GI tract including liver and kidney and reproduction organs (including breast for women and prostate for men)
Long-term effect - surgical procedures | 5, 10 and 20 years after randomisation
  1. Proportion of participants with any surgical procedure related to bariatric surgery: revisional surgery for late complications eg internal hernia, stomal ulcer; and conversion surgery eg change of operation from index procedure to another for weight regain or complications; or new bariatric procedures
  2. Proportion of participants with surgical procedures related to obesity and/or weight loss: eg cholecystectomy, body contouring surgery, elective arthroplasty
Long-term effect - fracture risk | 5, 10 and 20 years after randomisation
  1. Proportion of participants with any fracture
  2. Proportion of participants with major osteoporotic fracture (hip, spine, wrist, humerus)
Long-term effect - health economic and labour market attachment, employment status | 5, 10 and 20 years after randomisation
  Employment status each participant
Long-term effect - health economic and labour market attachment, salary | 5, 10 and 20 years after randomisation
  Salary for each participant
Long-term effect - health economic and labour market attachment, absence | 5, 10 and 20 years after randomisation
  Number of absence days
Long-term effect - health economic and labour market attachment, sick leave | 5, 10 and 20 years after randomisation
  Proportion of participants with any sick leave
Long-term effect - health economic and labour market attachment, long-term sick leave | 5, 10 and 20 years after randomisation
  Proportion of participants with long-term sick leave (more than 4 weeks continuous sickness absence)

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Dirksen, Ass Professor, Study Chair — Department of Medicine, Copenhagen University Hospital - Amager and Hvidovre
Locations (10):
- Denmark (4):
  - Steno Diabetes Center Aarhus, Aarhus Universitets Hospital, Aarhus
  - The Department of Medicine and Department of Surgery, University Hospital of South West Jutland, Esbjerg
  - The Department of Medicine and the Gastro Unit, Copenhagen University Hospital - Amager and Hvidovre, Hvidovre
  - Department of Surgery, Viborg Regional Hospital, Viborg
- United Kingdom (6):
  - St Richard's Hospital, Chichester, Sussex
  - Hartlands Hospital, University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Southmead Hospital, North Bristol NHS Trust, Bristol
  - The Whittington Hospital, London
  - Sunderland Royal Hospital, Sunderland
  - Musgrove Park Hospital, Somerset Foundation NHS Trust, Taunton

IPD SHARING:
Plan to Share IPD: Yes
After the results have been published, we aim to make a depersonalised dataset publicly available on e.g. ClinicalTrials.gov and/or the European Union (EU) Zenodo database (https://zenodo.org/). The final choice will reflect which platform(s) that are compliant with current legislation at that time.
Supporting Information: Study Protocol, SAP
Time Frame: When the results have been published
Access Criteria: Researchers with a protocol for their planned study

REFERENCES:
- [Derived] Tomova-Olsen SA, Kousgaard MB, Jensen KT, Reventlow S, Christiansen AL, Bojsen-Moller KN, Dirksen C, Overbeck G. Time, money, and weight loss: a qualitative study exploring patients' perspectives on randomization for bariatric surgery vs. an intensive non-surgical weight loss program. Trials. 2025 Apr 4;26(1):121. doi: 10.1186/s13063-025-08816-8. PMID 40186310
- See also: LightCOM website — https://www.regionh.dk/lightcom/uk/Pages/default.aspx